CLINICAL TRIAL: NCT07170943
Title: The Effect of Blueberry Supplementation on Cognitive Functioning in Older Adults
Acronym: BrainBerries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: too time-lengthy administrative process nationally - study no longer fits in PhD trajectory window
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Lisette de Groot, Dr., Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL77025.091.21
Record Dates: First submitted 2021-08-26; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Decline; Cognition Disorders in Old Age; Aging
Keywords: Cognition; Blueberry; Anthocyanins; Ageing
MeSH Terms: conditions — Cognitive Dysfunction | interventions — blueberry extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment is only partly masked for the participants; blueberry freeze-dried powder and placebo treatments are masked, but whole berry treatment is not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Whole blueberries (Experimental): Participants will consume a daily dose of 150g of whole blueberries
  Interventions: Other: Blueberry
- Freeze-dried blueberry powder (Experimental): Participants will consume a daily dose of 24g freeze-dried blueberry powder, equivalent to 150g whole blueberries
  Interventions: Dietary Supplement: Freeze-dried blueberry powder
- Placebo powder (Placebo Comparator): Participants will consume a daily dose of 24g colour- and flavour-matched maltodextrin powder
  Interventions: Dietary Supplement: Placebo powder

INTERVENTIONS:
Other: Blueberry — Daily consumption of blueberries
  Arms: Whole blueberries
Dietary Supplement: Freeze-dried blueberry powder — Daily consumption of a freeze-dried blueberry powder
  Arms: Freeze-dried blueberry powder
Dietary Supplement: Placebo powder — Daily consumption of a placebo powder
  Arms: Placebo powder

SUMMARY:
In this randomized placebo controlled intervention study, the effect of 12 weeks of supplementation with either 150g whole blueberries, freeze-dried blueberry powder (dose equivalent to 150g berries) versus placebo on cognitive functioning will be investigated in older adults.

DETAILED DESCRIPTION:
Dementia is a public health priority. The prevalence of dementia is rapidly increasing due to population ageing, posing a great social and economic impact on caregivers, families and society. This, in combination with the lack of effective treatment options, demonstrates the urgent need for better understanding on how to prevent and slow down progression of this condition. As ageing and dementia are associated with increased levels of inflammation, nutritional compounds that exhibit anti-inflammatory properties may propose a solution. Blueberries, a good source of anthocyanins, have shown anti-inflammatory properties in several human trials. Therefore, in this randomized placebo controlled intervention study, we aim to investigate the effect of 12 weeks of supplementation with either 150g whole blueberries or freeze-dried blueberry powder (dose equivalent to 150g berries) versus placebo on cognitive functioning in overweight older adults with mild memory complaints. Secondary objectives include the assessment of whole blueberry and freeze-dried blueberry powder supplementation on inflammatory markers, oxidative stress, intestinal health markers, vascular and metabolic health markers, mental well-being, and levels of neurotransmitters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65y
* Overweight, body mass index ≥25 kg/m2
* Mild memory complaints, i.e. ≥22 points on the Cognitive Failure Questionnaire (CFQ) and reporting to have memory complaints and being hampered by these complaints
* No mild cognitive impairment, i.e. ≥26 points on the Montreal Cognitive Assessment (MoCA)
* Able to understand and perform the study procedures

Exclusion Criteria:

* Body Mass Index (BMI) ≥35 kg/m2
* Current use of >500 mg/day of acetylsalicylic acid
* Current use of antidepressants
* Current use of medication that affects inflammation (anti-inflammatory medication)
* Current or recent (<1 month) use of berry supplements
* Current or recent (<1 month) use of anti-inflammatory dietary supplements such as fish oil, quercetin, curcumin, resveratrol, and/or other flavonoids
* Current or recent (<3 month) use of antibiotics.
* Berry consumption of more than 1 serving (150g) per week
* Not willing to quit anthocyanin-rich product consumption during the study period
* Allergy to berries/salicylates
* Having a current disease which interferes with the effect of berries/ freeze-dried berry powder and/or with the outcome measure (cognitive functioning), including diagnosis of dementia, psychiatric disorders, gastro-intestinal disease, diabetes, and cancer, as judged by a medical doctor
* Excessive alcohol consumption (on average >21 glasses/week for men and >14 glasses/week for women)
* Current participation in other scientific research

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Verbal fluency | 12 weeks
  Performance on verbal fluency

SECONDARY OUTCOMES:
Cognitive functioning | 12 weeks
  Rey Auditory Verbal Learning Test (RAVLT)
Cognitive function | 12 weeks
  Wechsler Digit Span Task (forward, backward, sequencing) WAIS-IV
Cognition | 12 weeks
  Symbol digit modalities test
Cognition | 12 weeks
  Trail Making Test (TMT) version A and B
Cognition | 12 weeks
  Stroop Color-Word test
Inflammation - CRP | 12 weeks
  Inflammatory blood marker: C-reactive protein
Inflammation - TNFalpha | 12 weeks
  tumor necrosis factor-alpha
Inflammation - IL6 | 12 weeks
  interleukin-6
Oxidative stress | 12 weeks
  total plasma nitric oxide (NO)
Oxidative stress | 12 weeks
  serum superoxide dismutase (SOD)
Intestinal health | 12 weeks
  Intestinal health markers as measured in blood and feces (microbiota composition, inflammatory fecal markers, microbiota-derived bioactive compounds, intestinal integrity markers
Metabolic health | 12 weeks
  Blood markers of metabolic health: plasma fasting glucose,
Metabolic health | 12 weeks
  Blood markers of metabolic health (plasma fasting glucose, Hb1Ac, triglyceride, adiponectin)
Metabolic health | 12 weeks
  Blood markers of metabolic health: Hb1Ac,
Metabolic health | 12 weeks
  Blood markers of metabolic health: triglyceride
Metabolic health | 12 weeks
  Blood markers of metabolic health: adiponectin
Mental well-being | 12 weeks
  Score on 12-item short form health survey
Mental well-being | 12 weeks
  profiles of mood states-short form (POMS)
Neurotransmitters | 12 weeks
  Levels of plasma neurotransmitters (dopamine, serotonin, (nor)adrenaline, and their metabolites)
Vascular health | 12 weeks
  Markers of vascular health (systolic blood pressure, diastolic blood pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, prof, Principal Investigator — Division of Human Nutrition and Health, Wageningen University and Research, The Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Starting 12 months after article publication. Sharing only upon reasonable request in consultation with the study team.
Time Frame: Starting 12 months after article publication.
Access Criteria: Upon reasonable request. Sharing will be done in consultation with the study team